CLINICAL TRIAL: NCT03239015
Title: Efficacy and Safety of Precision Therapy in Refractory Tumor (Long March Pathway)
Brief Title: Efficacy and Safety of Precision Therapy in Refractory Tumor
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Baodong Qin (Other)
Responsible Party: Sponsor-Investigator, Baodong Qin, Clinical Professor, Shanghai Changzheng Hospital
Organization: Shanghai Changzheng Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: Long March Pathway
Record Dates: First submitted 2017-07-28; First posted 2017-08-03 (Actual); Last update posted 2022-03-04 (Actual); Status verified 2022-02

CONDITIONS: Rare Tumor; Refractory Tumor
MeSH Terms: conditions — Neoplasms | interventions — Gefitinib; Erlotinib Hydrochloride; Afatinib; Trastuzumab; oxazolidine; olaparib; Everolimus; cabozantinib; Vemurafenib; dabrafenib; palbociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Targeted Drug Therapy Group (Experimental): All recruited patients with druggable molecular event will be treated with corresponding targeted drug including Gefitinib/Erlotinib/Afatinib, Trastuzumab, Oxazolidine, Olaparib, Everolimus, Cabozantinib, Vemurafenib/Dabrafenib, and Palbociclib. If no durggable target, PD-1/L1 inhibitor plus anti-angiogenic agent was used.
  Interventions: Drug: Gefitinib; Drug: Erlotinib; Drug: Afatinib; Drug: Trastuzumab; Drug: Oxazolidine; Drug: Olaparib; Drug: Everolimus; Drug: Cabozantinib; Drug: Vemurafenib; Drug: Dabrafenib; Drug: Palbociclib; Drug: PD-1/L1 inhibitor plus anti-angiogenic agent

INTERVENTIONS:
Drug: Gefitinib — Gefitinib is an FDA/CFDA approved targeted drugs used for EGFR mutation based on NGS results.
Drug: Erlotinib — Erlotinib is an FDA/CFDA approved targeted drugs used for EGFR mutation based on NGS results.
Drug: Afatinib — Afatinib is an FDA/CFDA approved targeted drugs used for EGFR mutation based on NGS results.
Drug: Trastuzumab — Trastuzumab is an FDA/CFDA approved targeted drugs used for Her2 amplification based on NGS results.
Drug: Oxazolidine — Oxazolidine is an FDA/CFDA approved targeted drugs used for ALK or ROS-1 or MET fusion based on NGS results.
Drug: Olaparib — Olaparib is an FDA/CFDA approved targeted drugs used for BRCA1/2 mutation based on NGS results.
Drug: Everolimus — Everolimus is an FDA/CFDA approved targeted drugs used for mTOR or PI3KCA mutation based on NGS results.
Drug: Cabozantinib — Cabozantinib is an FDA/CFDA approved targeted drugs used for RET mutation based on NGS results.
Drug: Vemurafenib — Vemurafenib is an FDA/CFDA approved targeted drugs used for BRAF mutation based on NGS results.
Drug: Dabrafenib — Dabrafenib is an FDA/CFDA approved targeted drugs used for BRAF mutation based on NGS results.
Drug: Palbociclib — Palbociclib is an FDA/CFDA approved targeted drugs used for CDK4/6 mutation or amplification based on NGS results.
Drug: PD-1/L1 inhibitor plus anti-angiogenic agent — PD-1/L1 inhibitor plus anti-angiogenic agent is a regimen used for refractory tumor without druggable target

SUMMARY:
This study is intended to evaluate efficacy and safety of targeted precision therapy in patients with refractory tumor, including rare tumor without standard recommended treatment and common tumor after multiple line of therapy.

DETAILED DESCRIPTION:
The individuals recruited in the present study are with solid tumor, mainly including two parts: first, rare tumor without standard recommended treatment such as atypical fibrous histiocytoma; second, common tumor after multiple line of therapy such as lung cancer, gastric cancer, colorectal cancer, etc. All patients have no any standard therapy based on NCCN guideline when recruiting. Next-generation sequence was used to detect druggable molecular event including gene mutation, gene fusion, amplification, etc. Then patients with molecular events were treated with corresponding targeted drug and followed-up, and not limited tumor type. PD-1/L1 inhibior plus anti-angiogenic agent was used in patients without durgguable targets. The efficacy and safety of these regimens were evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Malignant solid tumors diagnosed histologically;
* Common solid tumor patients have no any standard choice after multiple line of therapy; Rare solid tumor did not have any standard recommended treatment;
* Expected survival ≥ 1 month;
* ECOG / PS score: 0-2, and the main organ function to meet the following criteria: HB ≥ 90g / L, ANC ≥ 1.5 × 109 / L, PLT ≥ 80 × 109 / L,BIL <1.5 times the upper limit of normal (ULN); Liver ALT and AST <2.5 × ULN and if liver metastases, ALT and AST <5 × ULN; Serum Cr ≤ 1 × ULN, endogenous creatinine clearance ≥50ml/min

Exclusion Criteria:

* Patient still has standard treatment therapy based on NCCN guidance;
* Patient can not comply with research program requirements or follow-up;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 300 (Estimated)
Dates: Start 2017-01-01 (Actual); Primary Completion 2023-06-30 (Estimated); Study Completion 2023-12-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Evaluation of tumor burden based on RECIST criteria through study completion, an average of 2 months
  Proportion of patients with reduction in tumor burden of a predefined amount, including complete remission and partial remission

SECONDARY OUTCOMES:
Progress Free Survival | Evaluation of tumor burden based on RECIST criteria until first documented progress through study completion, an average of 2 months
  Time from treatment beginning until disease progression
Overall Survival | From date of treatment beginning until the date of death from any cause, through study completion, an average of 1 months
  Time from treatment beginning until death from any cause
Adverse Effect | Through study completion, an average of 1 months
  Incidence of Treatment-related adverse Events

CONTACTS AND LOCATIONS:
Overall Officials: Yuan-Sheng Zang, MD.PHD, Principal Investigator — Shanghai Changzheng Hospital
Locations (1):
- Shanghai Changzheng Hospital, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Qin BD, Jiao XD, Wang Z, Liu K, Wu Y, Ling Y, Chen SQ, Zhong X, Duan XP, Qin WX, Xue L, Guo ZH, Zang YS. Pan-cancer efficacy and safety of anlotinib plus PD-1 inhibitor in refractory solid tumor: A single-arm, open-label, phase II trial. Int J Cancer. 2023 Aug 15;153(4):815-825. doi: 10.1002/ijc.34546. Epub 2023 May 8. PMID 37155342
- [Derived] Jiao XD, Qin BD, Wang Z, Liu K, Wu Y, Ling Y, Qin WX, Wang MM, Yuan LY, Barreto SG, Kim AW, Mak K, Li H, Xu YY, Qiu XM, Wu M, Jin M, Xu LC, Zhong Y, Yang H, Chen XQ, Zeng Y, Shi J, Zhu WY, Ding QQ, Jia W, Liu SF, Zhou JJ, Shen H, Yao SH, Guo ZJ, Li T, Zhou PJ, Dong XW, Lu WF, Coleman RL, Akce M, Akladios C, Puccetti F, Zang YS. Targeted therapy for intractable cancer on the basis of molecular profiles: An open-label, phase II basket trial (Long March Pathway). Front Oncol. 2023 Feb 23;13:860711. doi: 10.3389/fonc.2023.860711. eCollection 2023. PMID 36910668